# UAB IRB Approved 10-Feb-2021 until 09-Feb-2022

#### **CONSENT FORM**

TITLE OF RESEARCH:

Comparative Effectiveness Trial Between a Clinic- and Complementary and Alternative Medicine Telerehabilitation Intervention for Adults with Multiple

Sclerosis

**IRB PROTOCOL:** IRB-161017003

**UAB PRINCIPAL** James Rimmer, Ph.D.

**INVESTIGATOR:** 

**SPONSOR:** The Patient-Centered Outcomes Research Institute (PCORI)

| General Information | You are being asked to take part in a research study. This research is voluntary, meaning you do not have to take part in it. The procedures, risks, and benefits are fully described further in the consent form. |
|---|---|
| Purpose | The purpose of this study is to solicit therapist opinions on the TEAMS Study program and its features (e.g., what they liked and disliked) to inform further refinements to the program. |
| Duration & Visits | You will be asked to complete a program satisfaction survey via email or mail, depending on your preference. This survey should take approximately 5 minutes to complete. You will also be asked to complete a 10-15 minute program satisfaction interview with research staff via phone or in person, depending on your preference. |
| Overview of Procedures | After the informed consent process, you will be asked to complete the brief program satisfaction interview and the survey, along with a demographic questionnaire. |
| Risks | There is a risk associated with potential loss of confidentiality. |
| Benefits | Your participation may provide valuable information to the medical community about remote exercise programs for adults with multiple sclerosis. |
| Alternatives | Your alternative is to not participate in this study. |

# **Purpose of the Research Study**

We are asking you to take part in a research study. The purpose of this study is to solicit TEAMS Study therapists' opinions on the TEAMS Study program and its features (e.g., what they liked and disliked) to inform further refinements to the program. This study will enroll TEAMS Study therapists across 43 TEAMS clinical sites in Alabama, Mississippi, and Tennessee. If you agree to participate in the study, you will be contacted for a brief interview, and/ or survey. This feedback will help study investigators continue to improve the program.

#### **Study Participation and Procedures**

Participants will be contacted by research staff and provided detailed information about the study procedures. If you agree to participate in the study, you will be asked to complete a program satisfaction survey, along with a demographic questionnaire, and an interview about your perceptions of the TEAMS Study program, such as


what you liked and disliked about the program. The survey will take approximately 5 minutes to complete,

#### **Alternatives**

Your alternative is to not participate in this study.

## **Confidentiality**

Information obtained about you for this study will be kept confidential to the extent allowed by law. However, research information that identifies you may be shared with the UAB Institutional Review Board (IRB) and other who are responsible for ensuring compliance with laws and regulation related to research, including people on behalf of Lakeshore Foundation, UAB School of Health Professions, and the Patient-Centered Outcomes Research Institute (PCORI, the funding agency), and the Office for Human Research Protections (OHRP).

The results of the study may be published for scientific purposes. These results could include your responses to surveys and/ or interviews. However, your identity will not be given out.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This web site will not include information that can identify you. At most, the web site will include a summary of the results. You can search this web site at any time.

### **Voluntary Participation and Withdrawal**

Whether or not you take part in this study is your choice. There will be no penalty if you decide


not to be in the study. If you decide not to be in the study, you will not lose any benefits you are otherwise owed. You are free to withdraw from this research study at any time. Your choice to leave the study will not affect your relationship with the clinic, Lakeshore Foundation or UAB.

If you are a UAB student, UAB employee, Lakeshore employee, or employee at this clinical site, taking part in this research is not a part of your class or work duties. You can refuse to enroll, or withdraw after enrolling at any time before the study is over, with no effect on your class standing, grades, or job at UAB, Lakeshore, or the clinic. You will not be offered or receive any special consideration if you take part in this research.

# **Cost of Participation**

There will be no cost to you for taking part in this study.

# Questions

If you have any questions, concerns, or complaints about the research, you may contact Dr. James Rimmer, He will be glad to answer any of your questions. Dr. Rimmer's number is (205) 975-9010.

If you have any questions about your rights as a research participant, or concerns or complaints about the research, you may contact the UAB Office of the IRB (OIRB) at (205) 934-3789 or toll free at 1-855-860-3789. Regular hours for the OIRB are 8:00 a.m. to 5:00 p.m. CT, Monday through Friday. You may also call this number in the event the research staff cannot be reached or you wish to talk to someone else.

### Legal Rights

You are not waiving any of your legal rights by signing this informed consent document.

#### **Use of Email Communications**

With your permission, the research team may use unencrypted emails to contact you regarding scheduling surveys and/ or interviews, or updates to information. Health information will not be emailed and you should not use email for any communication regarding health issues. There is a potential risk of loss of confidentiality when communicating via email. Unencrypted email communication is considered a non-secure method of sharing information. There is no guarantee that such communication (and any data associated with it) is private and will only be viewed by the intended recipient. By using unencrypted email, you acknowledge and accept this risk.

| monute respectively some simulations and accept time result |
|-------------------------------------------------------------|
| Please initial your choice below: |
| I would like to communicate via email. |
| I do not wish to communicate via email. |
| Signatures |

Your signature below indicates that you have read (or been read) the information provided above and agree to participate in this study. You will receive a copy of this signed consent form.


| Signature of Participant | Date |
|---------------------------------------|------|
| Signature of Person Obtaining Consent | Date |

